CLINICAL TRIAL: NCT05621850
Title: Impact of CErebral Endovascular PROcedures on the Systemic Immune responSe Response
Acronym: PROCESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 87RI22_0030 (PROCESS)
Record Dates: First submitted 2022-10-28; First posted 2022-11-18 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Arterio-venous Malformation
Keywords: Arterio-venous malformation; DMSO; Immune response; Cytokines
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cerebral AVM embolization (Experimental)
  Interventions: Other: Blood sample
- cerebral aneurism embolization (Other)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Based on supplementary blood sampled before embolization procedure and 6 hours and 24 hours after we will be analyzed cytokines concentration (Elisa test) and cortisol

SUMMARY:
In our ICU, it could notice that patients with cerebral arterio-venous malformation (AVM) treated with embolization develop more severe Ventilator Associated Pneumoniae (VAP) compare to other patients hospitalized for neurological diseases. The Dimethylsulfoxyde (DMSO), the solvent of the embolization implant, is known to have immune effect on vitro analysis. The investigator want to prove that exposition to embolization implant for a cerebral AMV modify the cytokines production involved the system immune's regulation.

DETAILED DESCRIPTION:
Cerebral AVM are defined by abnormal connections between arteries and veins. For treatment of this vascular malformation, embolization is the gold standard. Embolization agent is made with vinylic alcohol ethylene (EVOH) copolymer which (the embolization implant) and the DMSO which is the solvent. During the injection of the product, DMSO dissipates in the bloodstream, and the EVOH precipitates and forms the embolus. It knows that DMSO had in-vitro immune effect (inhibits signalizations ways of innate and acquired immune response, decrease of pro-inflammatory cytokines production and decrease INF-γ and TNF-α production). DMSO could decrease activation and recruitment of leukocytes, which could expose patients to an increased risk of infection.

The investigator will dose cytokines in 3 blood samples (preoperative, H+6 and H+24) in planned patient's hospitalized for cerebral AVM embolization. The cytokine content of the plasmas will be analyzed with multiplex ELISA technic

ELIGIBILITY:
Inclusion Criteria:

* Adult hospitalized for a planned cerebral embolization

Exclusion Criteria:

* Immunosuppressed patient or immunosuppressive treatment (corticosteroid included)
* Patient with auto-immune disease
* Hospitalization in ICU or for a planned or emergency surgery in the past three months
* Hospitalization for an active infection in the past three months
* Pregnancy
* Patients requiring steroid therapy to prevent postoperative nausea and/or vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Change in blood concentrations of cytokines of the innate immune response | Hour 0 and Hour 6
  Compare blood concentrations of cytokines (IL-1N, IL-10, IL-12p70, IL-6, IL-2, IL-4, IL-17A; TNF-a, TGF-b1, IFN-g) of the innate immune response between patients who underwent a cerebral AVM embolization procedure with patients who underwent a cerebral aneurysm embolization procedure between the expected peak at H6 and H0

SECONDARY OUTCOMES:
blood concentrations of cytokines of adaptive and innate immune response | Hour 0 and Hour 24
  Compare blood concentrations of cytokines (IL-1N, IL-10, IL-12p70, IL-6, IL-2, IL-4, IL-17A; TNF-a, TGF-b1, IFN-g) of adaptive and innate immune response between patients with cerebral AVM embolization procedures and brain aneurysms embolization
blood concentrations of cytokines | Hour 6
  Compare blood concentrations of cytokines (IL-1N, IL-10, IL-12p70, IL-6, IL-2, IL-4, IL-17A; TNF-a, TGF-b1, IFN-g)according to the duration of the embolization procedure at H6
blood concentrations of cytokines of adaptive immune response | Hour 0 and Hour 6
  Compare blood concentrations of cytokines (IL-1N, IL-10, IL-12p70, IL-6, IL-2, IL-4, IL-17A; TNF-a, TGF-b1, IFN-g)of adaptive immune response between patients with cerebral AVM embolization procedures and brain aneurysms embolization between the expected peak at H6 and H0
blood concentrations of cytokines according to the volume of embolizing agent | Hour 0 and Hour 6
  Compare blood concentrations of cytokines (IL-1N, IL-10, IL-12p70, IL-6, IL-2, IL-4, IL-17A; TNF-a, TGF-b1, IFN-g)according to the volume of embolizing agent
blood concentrations of cytokines according to the embolizing agent | Hour 0 and Hour 6
  Compare blood concentrations of cytokines (IL-1N, IL-10, IL-12p70, IL-6, IL-2, IL-4, IL-17A; TNF-a, TGF-b1, IFN-g)according to the embolizing agent used during the procedure
Cortisol production | Hour 0 and Hour 6
  Comparison of cortisol levels before and after AMV embolization procedure
lymphocyte subpopulations differences | Hour 24 and Hour 0
  Measurement of differences in lymphocyte subpopulations in patients with cAVM embolization procedure and cerebral aneurysm between the expected peak H24 and H0 in 10 patients in each arm

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No